CLINICAL TRIAL: NCT00482807
Title: Phase I Study Evaluating Extended Field Intensity Modulated Radiation Therapy and Docetaxel in Patients With Prostate Cancer Associated With Pelvic Node Metastasis
Brief Title: Radiation Therapy, Docetaxel, and Hormone Therapy in High-Risk Locally Advanced Metastasized Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0195-04-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Docetaxel; Goserelin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel, intensity-modulated radiation therapy and hormone therapy (Experimental): This phase I trial is studying the side effects and best dose of docetaxel when given together with intensity-modulated radiation therapy and hormone therapy in treating patients with high-risk locally advanced prostate cancer with pelvic lymph node metastasis.
  Interventions: Drug: bicalutamide; Drug: docetaxel; Drug: goserelin; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: bicalutamide
  Other Names: Casodex
Drug: docetaxel
  Other Names: Docefrez, Taxotere
Drug: goserelin
  Other Names: Zoladex
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high- dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as goserelin and bicalutamide, may lessen the amount of androgens made by the body. Giving radiation therapy together with chemotherapy and hormone therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel when given together with intensity-modulated radiation therapy and hormone therapy in treating patients with high-risk locally advanced prostate cancer with pelvic lymph node metastasis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine, preliminarily, the grade III or IV toxicity rate of concurrent extended-field intensity-modulated radiotherapy (IMRT), docetaxel, and androgen deprivation therapy in patients with high-risk, locally advanced prostate cancer with pelvic lymph node metastasis.

Secondary

* Determine, preliminarily, the progression-free survival of patients treated with this regimen.
* Determine the maximum tolerated dose of docetaxel when administered with concurrent IMRT in this patients.

OUTLINE: This is a dose-escalation study of docetaxel.

Patients receive combined androgen deprivation therapy (if not already on combined hormonal therapy) comprising goserelin acetate* subcutaneously once every 3 months for up to 2 years and oral bicalutamide once daily beginning on day 1 and continuing until the completion of radiotherapy. Beginning at approximately week 9 of androgen deprivation therapy, patients receive docetaxel IV over 1 hour once weekly for up to 9 weeks. Concurrently with chemotherapy, patients undergo intensity-modulated radiotherapy 5 days a week for up to 45 fractions (9 weeks).

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Note: *Not required for patients who have undergone bilateral orchiectomy

After completion of study therapy, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate

  o Locally advanced disease (T1 -T3b, N1 or N2, M0) at high risk for recurrence
  1. Biopsy-proven pelvic lymph node involvement
  2. No T4 lesion
* Prior androgen suppression within the past 14 months is allowed provided the following criterion is met:

  o No biochemical evidence of PSA progression after androgen withdrawal

  1. PSA progression, defined as 2 consecutive rising PSA values > 4.0 ng/mL taken ≥ 2 weeks apart
* Karnofsky performance status 80-100%
* absolute neutrophil count (ANC) ≥ 1,500/mm³
* Hemoglobin ≥ 10 g/dL
* Platelet count > 100,000/mm³
* Bilirubin normal
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* Meets 1 of the following criteria:
* Alkaline phosphatase (AP) normal and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 5 times upper limit of normal (ULN)
* AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
* AP ≤ 5 times ULN AND AST or ALT normal

Exclusion Criteria:

* No evidence of distant metastasis, including any of the following:

  * Bone metastasis
  * Pathologic or radiographic evidence of lymph node involvement above the L4 - L5 interspace
* No peripheral neuropathy > grade 1
* No significant comorbidity that would preclude radiotherapy
* No other prior malignancy except nonmelanoma skin cancer or any other cancer for which the patient has been disease-free for the past 5 years
* No hypersensitivity to docetaxel or other drugs formulated with polysorbate 80
* No history of Crohn's disease, ulcerative colitis, or irritable bowel syndrome
* No unrepaired inguinal hernia
* No prior pelvic or abdominal radiotherapy or prostate brachytherapy implant
* No prior prostatectomy
* No prior pelvic or abdominal surgery that resulted in excessive amounts of small intestine located within the pelvis
* No other concurrent investigational agents

Ages: 19 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-08-31 (Actual); Primary Completion 2010-03-09 (Actual); Study Completion 2010-03-09 (Actual)

PRIMARY OUTCOMES:
Toxicity rate | during therapy and follow-up, & for 5 years after radiation is completed
  Toxicity rate as assessed by NCI CTCAE v3.0

SECONDARY OUTCOMES:
Progression-free survival | From start of therapy up to 5 years after radiation is complete
  Time to Prostate Specific Antigen (PSA) failure
Maximum tolerated dose (MTD) of docetaxel | From start of therapy up to 5 years after radiation is complete
  Maximum tolerated dose (MTD) of docetaxel (dose below which excess dose limiting toxicity, DLT, observed.) If 3 patients treated at that dose, then added 3 should be entered, that process proceeds down, so MTD becomes highest dose where no more than 1 toxicity observed in 6 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hauke, MD, Principal Investigator — University of Nebraska; Elizabeth C Reed, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States